CLINICAL TRIAL: NCT03895437
Title: A Phase 2 Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of TOL-3021 in Patients With New Onset or Established Type 1 Diabetes Mellitus
Brief Title: Diabetes Autoimmunity Withdrawn In New Onset and In Established Patients
Acronym: SUNRISE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tolerion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOL-3021-231
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to treatment with TOL-3021 or placebo in a 2:1 fashion
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TOL-3021 (Experimental): TOL-3021 2 mg/mL
  Interventions: Biological: TOL-3021
- TOL-3021 Placebo (Placebo Comparator): TOL-3021 Placebo
  Interventions: Other: TOL-3021 Placebo

INTERVENTIONS:
Biological: TOL-3021 — TOL-3021 1 mg is a bacterial plasmid expression vector containing the coding sequences for the human proinsulin (hINS) gene.
  Arms: TOL-3021
Other: TOL-3021 Placebo — TOL-3021 Placebo
  Other Names: Placebo
  Arms: TOL-3021 Placebo

SUMMARY:
The study is a prospective, randomized, 52-week double-blind, placebo-controlled, multicenter trial in subjects with T1D followed by a 2-year safety follow-up.

DETAILED DESCRIPTION:
The SUNRISE study is a prospective, multi-center, double-blind, randomized, placebo-controlled trial in subjects aged 12.0 to <41.0 years diagnosed with T1D, as defined by American Diabetes Association (ADA) criteria, and within 5 years of diagnosis. Time of diagnosis is defined as the first day of insulin administration. Subjects will be stratified by duration (zero up to 1 year and 1 year up to five years) to ensure balance of disease duration across treatment and placebo groups in each strata. For analytical purposes, all subjects12-<41 will be considered cohort A, subjects aged 12-<18 will considered cohort B and subjects aged 18-<41 will be considered cohort C. For subjects aged 12-<18 (Cohort B), dosing will be staggered with an initial 6 subjects aged 14-<18 being enrolled with the last subject a having a minimum of 2 injections with at least 1 week follow-up after the 2nd injection. Safety data from this cohort will be evaluated before opening the study to subjects 12 and older. Subjects should be randomized no sooner than 6 weeks after diagnosis, unless glycemic range is adequately controlled as confirmed by time in glycemic range (70-180 mg/dL) >55% by CGM recording over 3 or more consecutive or non-consecutive days. Screening assessments will include a physical examination, a fundoscopic photograph, chemistry and hematology safety labs, urinalysis, 24-hour urine protein and creatinine, HbA1c, presence of T1D antibodies, and a 4-hour MMTT. Approximately 99 qualified subjects who meet all selection criteria will be randomized in a 2:1 ratio to treatment with TOL-3021 or placebo and treated for 52 weeks. Study drug treatments will be administered via an IM injection into a large muscle every week for 52 weeks. Continuous glucose monitoring (CGM) will be initiated within 5 days prior to the screening MMTT visit and continued through Week 52. Subjects will agree to diabetes management during the study with the goal of maintaining HbA1c levels of approximately 7.0% without frequent episodes of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 1 Diabetes Mellitus based on American Diabetes Association (ADA) criteria and within 5.0 years from diagnosis, defined as the first day of insulin administration.
2. Age at randomization of 12.0 - <41.0 years of age .
3. Adequate glycemic control as defined by HbA1c ≤7.9% based on point-of-care or local lab measurement and time in glycemic range (70-180 mg/dL) >55% by CGM recording over 3 or more consecutive or non-consecutive days within 5 days prior to baseline mixed meal tolerance test (MMTT).
4. On insulin therapy (total insulin dose >0.125 U/kg BW)
5. Presence of antibodies to at least one of the following antigens: GAD65, IA-2, ZnT8, or insulin if obtained within 10 days of the onset of exogenous insulin therapy, or documentation of positive antibodies. In the absence of a positive result for one of the specified antibodies, diagnosis of T1D as per the ADA guidelines..
6. Peak C-peptide during screening 4-hour mixed meal tolerance test (MMTT) ≥ 0.150 nmol/L.
7. Willingness to wear the Dexcom G6 continuous glucose monitoring (CGM) device and use according to instructions including recording of total daily insulin dose taken most of each day from screening to end of treatment period.
8. Written informed consent and, for subjects aged 12-<18 years of age, patient assent and parental or guardian consent, including authorization to release health information.
9. Willingness and ability of subject to comply with all study procedures of the study protocol, including attending all clinic visits.

Exclusion Criteria

1. Receiving a dose of acetaminophen >4,000 mg per day.
2. Body Mass Index (BMI) >32 kg/m² for patients 18 and older (>85th percentile for ages 12-17)
3. Previous immunotherapy for T1D within 2 years of enrollment.
4. Diagnosis of liver disease or hepatic enzymes, as defined by ALT and/or AST ≥ 2.5 times the upper limit of normal (ULN).
5. Hematology: white blood cells (WBC) <3 x 10⁹/L; platelets <100 x 10⁹/L; hemoglobin <10.0 g/dL. (Low WBC values may be repeated every 3-7 days, and results to be discussed with the Medical Monitor.) Any underlying conditions likely to impact red blood cell turnover.
6. Latent autoimmune diabetes of adults (LADA), which is generally associated with preceding history and treatment of T2D with medications typically used for treatment of T2D for more than 30 days.
7. Monogenic diabetes (MODY).
8. Estimated glomerular filtration rate (eGFR) <60 ml/min for ages 18-<41, and <75 ml/min per 1.73 m² for ages 12-<18.
9. History of malignancy, except for cancers in remission >5 years, or basal cell or in situ squamous cell carcinoma of the skin.
10. Significant cardiovascular disease (including inadequately controlled hypertension), history of myocardial infarction, unstable angina, use of anti-anginal medicines (e.g., nitroglycerin), or abnormal stress test, which, in the opinion of the Principal Investigator (PI), would interfere with participation in the trial.
11. Immunosuppressive therapy (systemic corticosteroids, cyclosporine, azathioprine, or biologics) within 30 days of screening.
12. Current or prior (within the last 30 days) use of metformin, sulfonylureas, glinides, thiazolidinediones, GLP1-RAs, DPP-IV inhibitors, pramlintide, or SGLT-2 inhibitors.
13. Current use of verapamil or α-methyldopa.
14. History of any organ transplant, including islet cell transplant.
15. Asthma that requires oral glucocorticoid therapy. Inhaled glucocorticoid therapy is permitted.
16. Active autoimmune or immune deficiency disorder including rheumatoid arthritis, moderate-to-severe psoriasis, inflammatory bowel disease, and other autoimmune conditions that may require treatment with TNF or other biologics. Permitted autoimmune disorders include T1D or well-controlled autoimmune conditions (e.g., thyroid disease, celiac disease, and sarcoidosis, all with stable non-immunosuppressive medications for the past 30 days).
17. Thyroid-stimulating hormone (TSH) at screening >7.5 mIU/L for ages 18-<41 years old and > 3.6mIU/L for ages 12-<18 years old. .
18. Adrenal insufficiency not adequately controlled with stable replacement glucocorticoid therapy.
19. Moderate non-proliferative retinopathy (NPDR) or proliferative retinopathy
20. Evidence of infection with HBV (as defined by hepatitis B surface antigen, HBsAg), HCV (anti-HCV antibodies), or HIV.
21. Subject is breastfeeding.
22. Positive urine pregnancy test at screening or at any time during the study (pregnancy tests must be performed as per the visit schedule). Females of childbearing potential must be excluded if they have a positive urine pregnancy test at screening or randomization or if they are not using medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, IUD, progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or 1 year or more postmenopausal must be specified in the subject's Case Report Form (CRF).
23. Males of reproductive potential who are unwilling to use medically acceptable birth control, unless the female partner is postmenopausal or surgically sterile.
24. Any social condition or medical condition that would, in the opinion of the PI, prevent complete participation in the study or would pose a significant hazard to the subject's participation.
25. Anticipated major surgery during the duration of the trial, which could interfere with participation in the trial.
26. History of drug or alcohol dependence within 12 months of screening.
27. Psychiatric disorder that would prevent subjects from giving informed consent.
28. Household members of current participants in this protocol.
29. Subjects who are not fluent in the English language.
30. Participation in other studies involving the administration of an investigational drug or experimental device, including the administration of an experimental agent for T1D within 30 days of screening, or use of an experimental therapeutic device for T1D within 30 days prior to screening. Subjects previously treated with diagnostic devices are not excluded.
31. Any current use of biotin or biotin containing supplements

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment effect on log-transformed MMTT C-peptide area under the curve (AUC) | 12. 16, 24 weeks
  The primary outcome is the TOL-3021 treatment effect as determined by a repeated measures analysis of change from baseline in the log-transformed MMTT C-peptide AUC at 12, 16, and 24 weeks

SECONDARY OUTCOMES:
Treatment effect on rates of clinically important hypoglycemia | 12, 24, 36, 52 weeks
  Rates of clinically important hypoglycemia events as defined by total measured glucose value of <54 mg/dL (3.0 mM/L) over each approximately 12-week period ending at Weeks 12, 24, 36, and 52 by a single blood glucose level, and by CGM, ≥10 consecutive minutes with glucose <54 mg/dL
Treatment effect on daily Insulin requirements | 24, 52 weeks
  Total daily insulin requirements in units per kilogram (kg) body weight
Treatment effect on HbA1c | baseline, 24, 52 weeks
  Change in HbA1c from baseline at Weeks 24 and 52
Treatment effect on log-transformed MMTT C-peptide area under the curve (AUC) | 12, 16, 24, 52 weeks
  Repeated measures analysis of change from baseline in the log-transformed MMTT C-peptide AUC at 12, 16, 24, and 52 weeks
Treatment effect on GCM measurement of glucose levels l< 70 and <55 mg/dL | 12, 16, 24, 52 weeks
  Number of times the CGM reports glucose levels of <70 and <55 mg/dL
Treatment effect on a Clinical responder analysis | 12, 16, 24, 52 weeks
  A clinical responder analysis defined as no change or an increase in C-peptide AUC from baseline between treatment and placebo at Weeks 12, 16, and 24 weeks. Upon completion of 52 week data, a similar analysis will include the 52 week data.
Treatment effect on non-fasting or fasting C-peptide single test | baseline, 12, 16, 24, 52 weeks
  Fasting or non-fasting C-peptide levels at baseline and at weeks 12, 16, 24, 52
Treatment effect on HbA1c | 52 weeks
  Proportion of subjects in each treatment arm with HbA1c levels <6.5% at Week 52
Treatment effect on CGM parameters | 12, 16, 24, 52
  Time in range of 70-180 mg/dL
Treatment effect on CGM parameters | 12, 16, 24, 52
  Time > 180 mg/dL;
Treatment effect on CGM parameters | 12, 16, 24, 52
  Time > 250 mg/dL
Treatment effect on CGM parameters | 12, 16, 24, 52
  Mean Glucose Coefficient of Variation
Treatment effect on CGM parameters | 12, 16, 24, 52
  Low Blood Glucose Index (LBGI)
Treatment effect on CGM parameters | 12, 16, 24, 52
  Glucose <70 mg/dL
Treatment effect on CGM parameters | 12, 16, 24, 52
  Area Under the Curve (AUC70)
Treatment effect on other measures of hypoglycemia | 12, 16, 24, 52 weeks
  Severe hypoglycemia (SH) events (impaired or loss of consciousness requiring assistance of another).
Treatment effect on other measures of hypoglycemia | 12, 16, 24, 52 weeks
  Documented symptomatic hypoglycemia (an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <70 mg/dl (3.9 mmol/L).
Treatment effect on other measures of hypoglycemia | 12, 16, 24, 52 weeks
  Total time <70 mg/dL by CGM.
Treatment effect on other measures of hypoglycemia | 12, 16, 24, 52 weeks
  Nocturnal hypoglycemia, i.e. severe or documented symptomatic episodes (as defined above) occurring after the subject has retired for the primary sleeping period.
Immunologic - Quantum dot (Q-dot) responses | at Week 52
  Quantum dot (Q-dot) responses within the qualifying subpopulation to confirm induction of specific autoantigen tolerance
Immunologic - Quantum dot (Q-dot) responses | at Week 52
  Comparison of quantum dot responses within the qualifying subpopulation to clinical outcomes to confirm correlation with specific autoantigen tolerance;
Immunologic - determine effect of treatment and predictive values of antibody response | at Week 52
  Regulatory/protective humoral immune response to proinsulin/insulin
Immunologic - determine effect of treatment and predictive values of antibody response | at Week 52
  Serum insulin autoantibody affinity for subjects
Immunologic - determine effect of treatment and predictive values of antibody response | at Week 52
  Insulin autoantibody isotypes (IgA and IgM) and IgG subclasses;;serum insulin, glutamic acid decarboxylase, IA-2, and ZnT8 antibodies by radio-binding assay (RBA) assay; competition assays of serum insulin and proinsulin IgM and IgG antibodies.
Immunologic - determine effect of treatment and predictive values of antibody response | at Week 52
  Serum insulin, glutamic acid decarboxylase, IA-2, and ZnT8 antibodies by radio-binding assay (RBA) assay
Immunologic - determine effect of treatment and predictive values of antibody response | at Week 52
  Competition assays of serum insulin and proinsulin IgM and IgG antibodies.
Safety Variables | 12, 16, 24, 52 weeks
  Clinical laboratory tests (hematology, chemistry, urinalysis)
Safety Variables | 12, 16, 24, 52 weeks
  Urine pregnancy test (UPT) for women of childbearing potential (WOCBP)c
Safety Variables | 12, 16, 24, 52 weeks
  Use of concomitant medications
Safety Variables | 12, 16, 24, 52 weeks
  Analysis of reported Adverse event (AEs)
Safety Variables | 12, 16, 24, 52 weeks
  Number of subjects with injection site reactions
Safety Variables | 12, 16, 24, 52 weeks
  Number of subjects with severe hypoglycemia or hyperglycemia events monitored by CGM
Events of Special Interest | 12, 16, 24, 52 weeks
  Number of subjects with systemic or hypersensitivity reactions associated with injection, which consist of fever, chills, headache, nausea, vomiting, and/or other signs and symptoms, such as anaphylaxis, wheezing dyspnea, urticaria, and hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fleming, M.D., Study Director — Tolerion, Inc.
Locations (23):
- United States (23):
  - Altman Clinical and Translational Research Institute UCSD, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Mills-Peninsula Medical Center, San Mateo, California
  - Stanford University, Stanford, California
  - Barbara Davis Center - University of Colorado Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - University of Miami Diabetes Research Institute, Miami, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - University of Iowa, Iowa City, Iowa
  - MedStar Health Research Institute, Baltimore, Maryland
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Joslin Diabetes Center- Adult & Pediatric, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Naomi Berrie Diabetes Center, Columbia University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - University of North Carolina Diabetes Care Center, Chapel Hill, North Carolina
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
We recognize that sharing anonymized data and other information from clinical trials can increase the speed and success of biomedical research in addressing unmet clinical need. We are following ongoing discussions among industry, the academic community, and other stakeholders regarding data sharing. Industry and its academic partners have not yet formulated a consensus on the amount, types, and forms of data that will be useful and beneficial to the public, or the process for sharing data. As a small, young company, we await the development of guidances and best practices for industry before issuing a comprehensive data sharing plan. For now, we defer a description of what data will be shared and the process for doing so. The protocol will be shared as part of study publication in a peer reviewed medical journal. The protocol will be available as a supplement to the publication and/or on the website of the publishing journal and upon request to the Sponsor (www.tolerion.bio)